CLINICAL TRIAL: NCT00113932
Title: UARK 2003-41: A Phase II Study of High-Dose Density Therapy With Tandem Autologous Transplants for Patients With Multiple Myeloma
Brief Title: UARK 2003-41: A Study of High-Dose Density Therapy in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2003-41
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Myeloma
Keywords: Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: High-Dose Density Therapy — Dexamethasone 40mg po 1-4, Thalidomide 200 mg po 1-6hrs then daily after transplant; Cisplatin* 10 mg/m2 Continuous infusion 1-4;Adriamycin 10 mg/m2 Continuous infusion 1-4;Cyclophosphamide 400 mg/m2 Continuous infusion 1-4; Etoposide 40 mg/m2 Continuous infusion 1-4; Pegfilgrastim 6 mg subcutaneously 6 and 13; Darbepoetin 200μg subcutaneously Between -6 to-1 +12, & every 2 weeks until HB >12 gm/dl***; Lovenox (or other LMWH) 40 mg subcutaneously Daily until Pltcount <30,000/μl

SUMMARY:
The purpose of this study is to find out if treating multiple myeloma (MM) patients with more intense chemotherapy and autologous transplant (high dose density therapy) early in the disease course will result in better treatment outcomes compared to patients treated in the past.

DETAILED DESCRIPTION:
This study will evaluate whether high-dose density treatment during the initial seven months, including tandem transplants within six months after starting therapy, results in superior event-free and overall survival rates as compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic multiple myeloma, previously treated or untreated.
* Patients previously untreated must not be eligible for UARK 2003-33.
* Karnofsky performance score > 60%, unless due to MM
* Patients must be <75 years of age at the time of registration
* Patient must not have had a prior auto- or allotransplant
* Patient must have signed an IRB-approved informed consent and understand the investigational nature of the study.
* Negative serology for HIV.
* Baseline studies within 60 days prior to registration; patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease. Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted. Patients unable to complete pulmonary function tests because of myeloma-related chest pain, must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.
* Patients with recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias are ineligible. Ejection fraction by ECHO or must be > 40% and must be performed within 60 days prior to registration, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the LVEF must be repeated.

Exclusion Criteria:

* Uncontrolled infection as defined in protocol section 5.1.11
* Liver function abnormalities with total bilirubin more than twice the upper limit of normal or AST or ALT more than three times the upper limit of normal
* Severe renal dysfunction, defined as a creatinine > 3mg/dl or a creatinine clearance of < 30ml/min
* Significant neurotoxicity, defined as grade > 2 neurotoxicity per NCI Common Toxicity Criteria
* Platelet count < 100,000/mm3, or ANC < 1,000/μl
* POEMS Syndrome
* Clinically significant hepatic dysfunction as noted by direct bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis
* New York Hospital Association (NYHA) Class III or Class IV heart failure
* Myocardial infarction within the last 6 months
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias
* Poorly controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Pregnant or potential for pregnancy. Women of childbearing potential will have a pregnancy [β-HCG] test at screening, and will be required to use a medically approved contraceptive method. Pregnancy testing will be performed prior to administration of each dose of study drug
* Breast-feeding women may not participate
* Prior adriamycin exposure >450 mg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-12; Primary Completion 2009-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate whether high-dose density treatment during the initial seven months, including tandem transplants within six months after starting therapy, results in superior event-free and overall survival rates as compared to historical controls. | seven months

SECONDARY OUTCOMES:
To evaluate the ability of pegfilgrastim to mobilize stem cells when administered following DTPACE in MM patients with active disease, compared to historical controls mobilized with DTPACE and either GM-CSF or G-CSF. | annually

CONTACTS AND LOCATIONS:
Overall Officials: Frits Van Rhee, MD, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States